CLINICAL TRIAL: NCT03933930
Title: Comparing the Prognosis of Lactate-directed and Goal-directed Therapy in Hyperthermic Intraperitoneal Chemotherapy.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patient wants to be recruited.
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, anchihhsu, Principal Investigator, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N201803039
Record Dates: First submitted 2019-04-12; First posted 2019-05-01 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Organ Failure, Multiple
MeSH Terms: conditions — Multiple Organ Failure | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactate-directed therapy (Experimental)
  Interventions: Other: Lactate-directed therapy; Other: Goal-directed therapy
- Goal-directed therapy (Experimental)
  Interventions: Other: Goal-directed therapy

INTERVENTIONS:
Other: Lactate-directed therapy — If the lactate level elevates, we transfuse pRBC to increase Hct>30%. If Hct >30%, dopamine infusion starts.
  Arms: Lactate-directed therapy
Other: Goal-directed therapy — If SVV>15%, transfuse lactate ringer/normal saline alternatively to keep SVV<15%.

SUMMARY:
Hyperthermic intraperitoneal chemotherapy is a major surgery for tumor peritoneal metastasis. For anesthesiologist, the intra-operative fluid control is always a big challenge. We try to compare the prognosis of lactate-directed and goal-directed therapy. We expect to confirm the better prognosis of lactate-directed therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* Unable to set arterial line Severe liver or renal disease Severe heart disease Unconscious patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-06 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
pulmonary complication | 1 week
  X-ray findings of airspace or interstitial opacity, lobar consolidation, or pleural effusions; severe respiratory failure requiring respiratory support

SECONDARY OUTCOMES:
Renal complication | 1 week
  oliguria with urine output<0.5 ml/kg/h for more than 4 h, creatinine increase>30 % of preoperative values, dialysis

IPD SHARING:
Plan to Share IPD: No